CLINICAL TRIAL: NCT02071953
Title: Clinical Evaluation of an Experimental Universal Adhesive Used With and Without Phosphoric Acid Pretreatment in Posterior Composite Resin Restorations
Brief Title: Comparative Study of Experimental Dental Adhesive With and Without Phosphoric Acid Pretreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply International (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 765-550; 815642 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2014-02-21; First posted 2014-02-26 (Estimated); Results first posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adhesive without acid pretreatment (Experimental): Experimental adhesive w/out phosphoric acid in post. rest.
  Interventions: Device: Experimental adhesive w/out phosphoric acid in post. rest.
- Adhesive with acid pretreatment (Active Comparator): Experimental adhesive with phosphoric acid in post. rest.
  Interventions: Device: Experimental adhesive with phosphoric acid in post. rest.

INTERVENTIONS:
Device: Experimental adhesive w/out phosphoric acid in post. rest. — Experimental adhesive without phosphoric acid in posterior restorations
  Arms: Adhesive without acid pretreatment
Device: Experimental adhesive with phosphoric acid in post. rest. — Experimental adhesive with phosphoric acid in posterior restorations
  Arms: Adhesive with acid pretreatment

SUMMARY:
The intent of this study is to evaluate the clinical performance of an experimental dental bonding agent for use with dental restorative composites with and without pretreatment of the tooth dentin and enamel using phosphoric acid etching.

DETAILED DESCRIPTION:
The intent of this study is to evaluate the clinical performance of an experimental dental bonding agent (adhesive) for use with dental restorative composites with and without pretreatment of the tooth dentin and enamel using phosphoric acid etching.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of Class I and Class II restorations in premolars and molars.

Exclusion Criteria:

* Patients with fewer than 20 teeth
* Patients exhibiting poor oral hygiene or uncontrolled periodontal disease
* Pregnant women or lactating mothers
* Patients with known allergies to HEMA or resin-based materials
* Patients with medical conditions that would contraindicate dental treatment
* Patients with xerostomia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Walter, DDS, Principal Investigator — University of Pennsylvania; Alan M. Atlas, DMD, Principal Investigator — Academy House of Professional Offices

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: teeth
Groups:
- Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration: Experimental adhesive without phosphoric acid in posterior restoration
- Experimental Adhesive w/ Phosphoric Acid in Post Restoration: Experimental adhesive with phosphoric acid in post restoration
Period: Overall Study
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration | Experimental Adhesive w/ Phosphoric Acid in Post Restoration
Started | 35; 53 teeth (Number of participants is being calculated more than once per row. Note that most participants had subject teeth in both arms of the study.) | 35; 54 teeth (Number of participants is being calculated more than once per row. Note that most participants had subject teeth in both arms of the study.)
Completed | 18; 30 teeth (Number of participants is being calculated more than once per row. Note that most participants had subject teeth in both arms of the study.) | 21; 34 teeth (Number of participants is being calculated more than once per row. Note that most participants had subject teeth in both arms of the study.)
Not Completed | 17; 23 teeth | 14; 20 teeth

BASELINE CHARACTERISTICS:
Population: Note: The units analyzed are teeth and most participants had more than one tooth treated in this study. A same participant could have individual teeth assigned to either arm. Most participants had teeth counted in both arms. A participant could have up to 4 units (teeth) treated and each unit was randomly assigned to one of the two arms.
  Participants were randomized to exclude bias due to age and sex.
Units Other Than Participants: teeth
Groups:
- Experimental: Adhesive With and Without Acid Pretreatment: Experimental adhesive with and without phosphoric acid in posterior restoration
Arm/Group | Experimental: Adhesive With and Without Acid Pretreatment
Number analyzed (Participants) | 37
Number analyzed (teeth) | 107
Age, Categorical [Count of Units; unit: teeth] — Patients were between 18 and 65 years of age. No additional information was recorded regarding patient age.
  teeth
    <=18 years | 0
    Between 18 and 65 years | 107
    >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 20
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Color Match
Description: The color match will be assessed clinically according to Ryge (1973)* for matching with adjacent teeth and stability of color matching over time.
  Assessments will be done to the following criteria:
  Alpha= Restoration matches adjacent tooth structure in shade and/or translucency.
  Bravo= Mismatch in shade and/or translucency is within normal range of tooth shades.
  Charlie= Mismatch in shade and/or translucency is outside normal range of tooth shades.
  *As per the Investigation Protocol, United States Public Health Service (USPHS) direct evaluation procedures were conducted using modified methods reported by Ryge in 1973.
  As described by Ryge in 1973, the term "clinical assessment" means a visual examination by a dentist, using a mouth mirror, an explorer, and supplementary lighting as needed.
Time Frame: Baseline, 6 months, 18 months; Note: The 36 month evaluation was an option in the protocol at the time of investigation initiation. The study was concluded at 18 months. Thus 36 month data does not exist.
Population: This is the total number of participants remaining at the end of the study who completed the 18 month follow-up. 22 participants presented for the 18 month evaluation. Most participants had subject teeth in both arms of the study. The reporting below is on the number of teeth, not subjects.
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Groups:
- Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline): Experimental adhesive without phosphoric acid in posterior restoration (Baseline)
- Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (Baseline): Experimental adhesive with phosphoric acid in posterior restoration (Baseline)
- Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (6-month): Experimental adhesive without phosphoric acid in posterior restoration (6-month)
- Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (6-month): Experimental adhesive with phosphoric acid in posterior restoration (6-month)
- Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month): Experimental adhesive without phosphoric acid in posterior restoration (18-month)
- Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month): Experimental adhesive with phosphoric acid in posterior restoration (18-month)
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month) | Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 18 | 21
Number analyzed (teeth) | 53 | 54 | 50 | 52 | 30 | 34
teeth
  Alpha | 53 | 54 | 50 | 52 | 30 | 34
  Bravo | 0 | 0 | 0 | 0 | 0 | 0
  Charlie | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Marginal Discoloration
Description: Marginal discoloration will be assessed clinically according to Ryge (1973)* over time.
  Assessments will be done to the following criteria:
  Alpha= No visual evidence of marginal discoloration. Bravo= Marginal discoloration present but has not penetrated in a pulpal direction.
  Charlie= Marginal discoloration has penetrated in a pulpal direction.
  *As per the Investigation Protocol, United States Public Health Service (USPHS) direct evaluation procedures were conducted using modified methods reported by Ryge in 1973.
  As described by Ryge in 1973, the term "clinical assessment" means a visual examination by a dentist, using a mouth mirror, an explorer, and supplementary lighting as needed.
Time Frame: Baseline, 6 months, 18 months. Note: The 36 month evaluation was an option in the protocol at the time of investigation initiation. The study was concluded at 18 months. Thus 36 month data does not exist.
Population: as for outcome 1
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Groups:
- Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline): For experimental adhesive without phosphoric acid in posterior region Arm (Baseline)
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month) | Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 18 | 21
Number analyzed (teeth) | 53 | 54 | 50 | 52 | 30 | 34
teeth
  Alpha | 53 | 54 | 50 | 52 | 27 | 34
  Bravo | 0 | 0 | 0 | 0 | 3 | 0
  Charlie | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Marginal Integrity
Description: Change in marginal integrity will be assessed clinically according to Ryge (1973)* over time.
  Assessments will be done to the following criteria:
  A= Explorer does not catch or slight catch with no visible crevice. B= Explorer catches and crevice is visible but no exposure of dentin or base. C= Explorer penetrates crevice and defect extended to amelo-dentinal junction. D= Restoration is fractured, mobile, or missing in part or in toto.
  *As per the Investigation Protocol, United States Public Health Service (USPHS) direct evaluation procedures were conducted using modified methods reported by Ryge in 1973.
  As described by Ryge in 1973, the term "clinical assessment" means a visual examination by a dentist, using a mouth mirror, an explorer, and supplementary lighting as needed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month) | Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 18 | 21
Number analyzed (teeth) | 53 | 54 | 50 | 52 | 30 | 34
teeth
  Alpha | 53 | 53 | 49 | 52 | 26 | 34
  Bravo | 0 | 0 | 0 | 0 | 3 | 0
  Charlie | 0 | 0 | 0 | 0 | 0 | 0
  Delta | 0 | 1 | 1 | 0 | 1 | 0

4. Primary Outcome: Presence of Secondary Dental Caries (Cavities)
Description: Change in presence of secondary dental caries will be assessed clinically according to Ryge (1973)* over time.
  Assessments will be done to the following criteria:
  A= No caries present. D= Caries present associated with the restoration.
  *As per the Investigation Protocol, United States Public Health Service (USPHS) direct evaluation procedures were conducted using modified methods reported by Ryge in 1973.
  As described by Ryge in 1973, the term "clinical assessment" means a visual examination by a dentist, using a mouth mirror, an explorer, and supplementary lighting as needed.
  Note: Secondary caries is a categorical, dichotomous variable, i.e. there is caries or not. This was assessed clinically and radiographically by a trained professional (dentist).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month) | Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 18 | 21
Number analyzed (teeth) | 53 | 54 | 50 | 52 | 30 | 34
teeth
  Alpha | 53 | 54 | 50 | 52 | 30 | 34
  Delta | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Presence of Restoration Fractures (Localized or Bulk)
Description: The restoration will be assessed clinically according to Ryge (1973)* for presence of fractures over time.
  Assessments will be done to the following criteria:
  A= Smooth restoration surface with no irregularities. B= Slightly rough or pitted restoration surface. Can be refinished. C= Deeply pitted or grooved (not related to anatomy) restoration finish. Can not be refinished.
  D= Restoration surface is fractured or flaking.
  *As per the Investigation Protocol, United States Public Health Service (USPHS) direct evaluation procedures were conducted using modified methods reported by Ryge in 1973.
  As described by Ryge in 1973, the term "clinical assessment" means a visual examination by a dentist, using a mouth mirror, an explorer, and supplementary lighting as needed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month) | Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 18 | 21
Number analyzed (teeth) | 53 | 54 | 50 | 52 | 30 | 34
teeth
  Alpha | 52 | 53 | 47 | 52 | 27 | 34
  Bravo | 0 | 0 | 2 | 0 | 2 | 0
  Charlie | 0 | 0 | 0 | 0 | 0 | 0
  Delta | 1 | 1 | 1 | 0 | 1 | 0

6. Primary Outcome: Post-operative Sensitivity
Description: Patient will be interviewed to assess post-operative sensitivity according to the following criteria:
  A= No sensitivity. B= Mild sensitivity. C= Moderate sensitivity with no restoration replacement required. D= Sever sensitivity. Replacement of restoration is required.
  Tooth sensitivity will be assessed at baseline and each follow-up appointment using cold thermal test (Endo-Ice, Hygienic) and Electric Pulp Test (EPT) when indicated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month) | Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 18 | 21
Number analyzed (teeth) | 53 | 54 | 50 | 52 | 30 | 34
teeth
  Alpha | 51 | 53 | 50 | 52 | 30 | 34
  Bravo | 2 | 0 | 0 | 0 | 0 | 0
  Charlie | 0 | 0 | 0 | 0 | 0 | 0
  Delta | 0 | 1 | 0 | 0 | 0 | 0

7. Primary Outcome: Surface Condition of Restoration
Description: The change in surface condition of restoration will be assessed clinically according to Ryge (1973)* over time.
  Assessments will be done to the following criteria:
  A= Restoration is continuous with existing anatomic form. B= Restoration is discontinuous with existing anatomic form but missing material is not sufficient to expose dentin or lining.
  C= Sufficient restorative material is lost to expose dentin.
  *As per the Investigation Protocol, United States Public Health Service (USPHS) direct evaluation procedures were conducted using modified methods reported by Ryge in 1973.
  As described by Ryge in 1973, the term "clinical assessment" means a visual examination by a dentist, using a mouth mirror, an explorer, and supplementary lighting as needed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (Baseline) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/ Phosphoric Acid in Posterior Restoration (6-month) | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month) | Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)
Number analyzed (Participants) | 18 | 35 | 34 | 34 | 18 | 21
Number analyzed (teeth) | 53 | 54 | 50 | 52 | 30 | 34
teeth
  AlphaB | 53 | 54 | 47 | 52 | 29 | 34
  Bravo | 0 | 0 | 3 | 0 | 1 | 0
  Charlie | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Gingival Inflammation Index
Description: Patient's gingiva will be assessed clinically according to Ryge (1973)* over time.
  Assessments will be done to the following criteria:
  0 = Normal gingiva.
  1. = Mild inflammation, slight change in color, slight edema, no bleeding upon probing.
  2. = Moderate inflammation, redness; edema and glazing; bleeding upon palpation.
  3. = Severe inflammation, marked redness and edema, ulceration, tendency to spontaneous bleeding.
     * As described by Ryge in 1973, the term "clinical assessment" means a visual examination by a dentist, using a mouth mirror, an explorer, and supplementary lighting as needed.
  Note: At 6 months data was not reported. At Baseline, all patients presented a score of 0. Any patient with a score greater than zero would have been excluded at baseline.
  Patients who received Class I restorations were not assessed as these restorations are limited to the chewing surface and not related to the health of gums.
Time Frame: 18 months; Note: The 36 month evaluation was an option in the protocol at the time of investigation initiation. The study was concluded at 18 months. Thus 36 month data does not exist.
Population: This is the total number of participants remaining at the end of the study who completed the 18 month follow-up. 22 participants presented for the 18 month evaluation. Most participants had subject teeth in both arms of the study. The reporting below is on the number of teeth, not subjects. Twenty-two (22) of the restorations were Class I and have no interaction with the gingival tissue and therefore were not scored. Scores below are for the remaining 42 Class II restorations.
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Groups:
- Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month)-Class II Restoration: Experimental adhesive w/out phosphoric acid in posterior restoration (18-month)-Class II restorations
- Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)-Class II Restoration: Experimental adhesive with phosphoric acid in posterior restoration (18-month)-Class II restorations
Arm/Group | Experimental Adhesive w/Out Phosphoric Acid in Posterior Restoration (18-month)-Class II Restoration | Experimental Adhesive w Phosphoric Acid in Posterior Restoration (18-month)-Class II Restoration
Number analyzed (Participants) | 18 | 21
Number analyzed (teeth) | 22 | 20
teeth
  0 | 12 | 9
  1 | 9 | 11
  2 | 1 | 0
  3 | 0 | 0

ADVERSE EVENTS:
Groups:
- Adverse Events: Intervention was the use of phosphoric acid. In the experimental group phosphoric acid was used. In the control group, phosphoric acid was not used.
  Dosage: As visually needed to cover exposed dentin and prepared enamel. Frequency: Once, at placement of filling
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No